CLINICAL TRIAL: NCT02307578
Title: An Extended Access Program (EAP) for Perampanel
Status: No longer available | Type: Expanded Access
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: E2007-G000-409
Record Dates: First submitted 2014-12-02; First posted 2014-12-04 (Estimated); Last update posted 2025-09-15 (Actual); Status verified 2025-03

CONDITIONS: Primary Generalized Tonic-Clonic or Partial Onset Seizures; Lennox Gastaut Syndrome
Keywords: Perampanel; Fycompa; Primary Generalized Tonic-Clonic Seizures; E2007-G000-332; E2007
MeSH Terms: conditions — Lennox Gastaut Syndrome | interventions — perampanel

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Perampanel — Perampanel will be available in 2-milligrams (mg), 4-mg and 8-mg tablets and as 0.5 milligram per milliliter (mg/mL) oral suspension. Participants will start this EAP with the dose that they were receiving at the end of their participation in Study E2007-G000-332, Study E2007-G000-311, E2007-G000-238, E2007-G000-338 or EAP E2007-G000-401. Doses of perampanel can be adjusted based on clinical judgment.
  Other Names: E2007, Fycompa

SUMMARY:
The main objective of this EAP is to ensure that participants participating in Study E2007-G000-332, Study E2007-G000-311, E2007-G000-238, E2007-G000-338 or EAP E2007-G000-401 continue to have access to perampanel until such time that the appropriate formulation of perampanel becomes commercially available in the country in which they reside or until no participants remain in the EAP.

ELIGIBILITY:
Inclusion criteria:

1. Participants who have completed their participation in Study E2007-G000-332, Study E2007-G000-311, E2007-G000-238, E2007-G000-338, or who are being rolled over from EAP E2007-G000-401 and, who in the opinion of the treating physician, continue to demonstrate a positive benefit-to-risk ratio from treatment with perampanel.
2. Participants who provide informed consent where applicable per local requirements.
3. Female participants of childbearing potential must agree for the duration of the program and for a period of at least 1 month following last dose of perampanel to be abstinent or to commit to the consistent and correct use of a medically acceptable method of birth control (example, a double-barrier method [condom plus spermicide, condom plus diaphragm with spermicide]).

Exclusion criteria:

1. Participants who reside in countries where the appropriate formulation of perampanel is commercially available.
2. Female participants who are nursing, pregnant, or planning to become pregnant.

Min Age: 1 Year | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (27):
- Belgium (3):
  - Cliniques Universitaires Saint-Luc, Brussels
  - Hôpital Universitaire des Enfants Reine Fabiola, Brussels
  - Centre Neurologique William Lennox, Ottignies
- Hospital Padre Hurtado, Santiago, Chile
- Czechia (2):
  - Artroscan, Ostrava-Trebovice
  - Všeobecná fakultní nemocnice, Pragtis s.r.o, Prague
- Estonia (2):
  - Oy Neurodiagnostika Ap, Tallinn
  - Tartu University Hospital, Tartu
- Hungary (7):
  - Dél-Pesti Centrumkórház Országos Hematológiai és Infektológiai Intézet, Budapest
  - Magyarorszagi Reformatus Egyhaz (MRE) Bethesda Gyermekkorhaza, Budapest
  - Országos Idegsebészeti Tudományos Intézet, Budapest
  - Rajna és Fiai Kereskedelmi és Szolgáltató Kft., Budapest
  - Servus Salvus Egeszsegugyi Szolgaltato Kft., Budapest
  - Borsod-Abaúj-Zemplén Megyei Központi Kórház és Egyetemi Oktató Kórház, Miskolc
  - Pécsi Tudományegyetem, Pécs
- Latvia (2):
  - Childrens University Hospital, Riga
  - Riga 1st Hospital, Riga
- Klaipeda University Hospital, Klaipėda, Lithuania
- Poland (5):
  - Uniwersyteckie Centrum Kliniczne - PPDS, Gdansk
  - Nzoz Novo-Med, Katowice
  - NZOZ Centrum Neurologii Dzieciecej i Leczenia Padaczki, Kielce
  - Szpital Kliniczny im. H.Swiecickiego Uniwersytetu Medycznego im. Karola Marcinkowskiego w Poznaniu, Poznan
  - Instytut Psychiatrii Neurologii, Warsaw
- Clinical Centre of Serbia, Belgrade, Serbia
- Spain (3):
  - Hospital Sant Joan de Deu, Esplugues de Llobregat
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Virgen del Rocio -, Seville